CLINICAL TRIAL: NCT02807129
Title: Fragmentation of Elastin as a Biological Marker of Frailty and Impact in Tumor Progression in Elderly Patients With Cancer
Acronym: AgElOn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PO12140
Record Dates: First submitted 2016-06-16; First posted 2016-06-21 (Estimated); Last update posted 2026-01-21 (Actual); Status verified 2025-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Urine Specimen Collection

ARMS (1):
- patients (Experimental)
  Interventions: Biological: blood withdrawn; Biological: urine collection

INTERVENTIONS:
Biological: blood withdrawn
Biological: urine collection

SUMMARY:
The aim of the study is to evaluate frailty in patients aged ≥ 65 years with cancer. The elderly population is very heterogeneous, it is necessary to evaluate these elderly patients before treatment to assess the risk-benefit balance. To date, this assessment relies on subjective clinical methods often not optimal, and slow to implement. An innovative method of evaluation could be the determination of elastin peptides. Indeed, the rate of these peptides, which are linked to serious conditions associated with age, rising inexorably with age and dose could help determine more objectively the type of treatment to offer older patients.

Expected results : This study will allow better identification of the group of frail elderly through more relevant biological marker that clinical assessment, often subjective and not available within a period compatible with the treatment of newly diagnosed cancer. This biological assessment will also enable optimal management of elderly patients in particular by allowing the geriatrician better efficiency.

ELIGIBILITY:
Inclusion Criteria:

* 65 years or older
* diagnosis of cancer
* affiliation to a social security scheme
* Signed informed consent for the study and for the collection of biological samples

Exclusion Criteria:

* Patient protected by law (guardianship, trusteeship)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 296 (Actual)
Dates: Start 2014-01-29 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2023-01-16 (Actual)

PRIMARY OUTCOMES:
elastin peptides quantification | up to 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France

REFERENCES:
- [Background] Salesse S, Odoul L, Chazee L, Garbar C, Duca L, Martiny L, Mahmoudi R, Debelle L. Elastin molecular aging promotes MDA-MB-231 breast cancer cell invasiveness. FEBS Open Bio. 2018 Aug 2;8(9):1395-1404. doi: 10.1002/2211-5463.12455. eCollection 2018 Sep. PMID 30186741